CLINICAL TRIAL: NCT02539199
Title: Vaginally Administered Versus Per Oral Misoprostol in Induction of Labour: a Randomized Trial
Brief Title: Vaginally Administered Versus Per Oral Misoprostol in Induction of Labour
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R15109M; 2015-001972-23 (EudraCT Number)
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Labour Induction
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol modified-release pessary (Active Comparator)
  Interventions: Drug: Misoprostol, modified-release pessary
- Misoprostol, per-oral tablets (Active Comparator)
  Interventions: Drug: Misoprostol, per-oral tablets

INTERVENTIONS:
Drug: Misoprostol, modified-release pessary — Misoprostol pessary (7 ug/h) placed in vaginal fornix until labour is induced or maximum 24 hours
  Other Names: Misodel
  Arms: Misoprostol modified-release pessary
Drug: Misoprostol, per-oral tablets — First day: 50 ug PO in every 4 hours maximum 3 times per day. Second day: 100 ug PO in every 4 hours maximum 3 times per day. Third day: 50 ug vaginally in every 4 hours maximum 3 times per day or until labour is induced.
  Other Names: Cytotec
  Arms: Misoprostol, per-oral tablets

SUMMARY:
The purpose of this study is to investigate the effectiveness and safety of vaginally administered misoprostol (Misodel) versus per orally administered misoprostol (Cytotec) in induction of labour in nulliparous women.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* Singleton at term pregnancy (>36+6 weeks)
* Unfavourable cervix (Bishop score < 6)
* Fetal cephalic position

Exclusion Criteria:

* Pre-term pregnancy (<37 weeks)
* Multiple pregnancy
* Rupture of membranes
* Other than fetal cephalic position
* Intra-uterine growth retardation
* Severe pre-eclampsia
* Severe hypertension
* Previous cesarean section

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2015-09; Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Cesarean section rate | at time of child birth

SECONDARY OUTCOMES:
The time from beginning of induction to child birth | up to child birth
Neonatal Apgar score | 1, 5, 10 minutes after child birth

CONTACTS AND LOCATIONS:
Overall Officials: Kati Tihtonen, PhD, MD, Principal Investigator — Tampere University Hospital
Locations (5):
- Finland (5):
  - Helsinki University hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku